CLINICAL TRIAL: NCT07052266
Title: Feasibility of Obstetric and Cancer Universal Screening
Brief Title: Trial of Combined Obstetric Carrier Screening and Hereditary Cancer Screening
Acronym: FOCUS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Myriad Genetics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 25-02028559
Record Dates: First submitted 2025-06-26; First posted 2025-07-04 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Hereditary Cancer Syndromes
Keywords: Genetic Testing; Carrier Screening; Prenatal Screening; Reproductive Genetic Testing; Feasibility Study; Universal Screening
MeSH Terms: conditions — Neoplastic Syndromes, Hereditary

STUDY DESIGN:
Intervention Model Description: The investigators are offering hereditary cancer screening genetic test to patients already receiving standard of care obstetric carrier screening.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Collection of HCS and OCS for patients receiving obstetrical-related care (Experimental): The first arm is for an obstetrical/prenatal (standard arm) setting
  Interventions: Genetic: MyRisk Hereditary Cancer Test
- Collection of HCS and OCS for patients receiving preconception/fertility care (Experimental): This second arm is at reproductive endocrinology and infertility clinics (preconception arm)
  Interventions: Genetic: MyRisk Hereditary Cancer Test

INTERVENTIONS:
Genetic: MyRisk Hereditary Cancer Test — Subjects that are planning to proceed with OCS and enrolled in the trial will be contacted by the genetics clinician (by telephone or in person, based on subject preference) to review the option for HCS in addition to OCS. The WCM genetics clinician will review the potential risks and benefits, possible findings, and implications of findings for HCS. The genetics clinician will follow WCM standards (outlined by the WCM Genetics and Personalized Cancer Prevention Program https://wcinyp.org/GPCP) for informed consent counseling on the potential risks/benefits of HCS. The counseling regarding OCS will have already been performed by the obstetrical team as part of the standard of care. The genetics clinician will review that OCS is being performed as part of the patient's standard of care prenatal visit and HCS is an additional component that is being performed as part of participation in this clinical trial.

SUMMARY:
The investigators hypothesize that pregnancy and preconception care may be a feasible and effective time to offer inherited cancer risk screening. This study will assess interest in cancer genetic testing among patients receiving routine prenatal or preconception/fertility care. The goal is to evaluate the acceptability of BRCA1/2 testing when offered alongside standard prenatal genetic screening. The study will also explore whether universal screening in this population could support early cancer prevention and be cost-effective, especially among underserved populations.

DETAILED DESCRIPTION:
The purpose of this study is to prospectively offer obstetric patients combined hereditary cancer screening (HCS) and obstetric carrier screening (OCS) to see if patients decide they want HCS in addition to their OCS. Preconception and pregnancy represent a unique window of opportunity for women to engage and interact with the healthcare system. With the proposed trial, the investigators aim to change the paradigm of obstetrical-related genetic testing to include potentially life-saving HCS.

Approximately 25% of the general population in the U.S. meets established criteria to recommend genetic counseling and testing for hereditary cancer syndromes, but less than 1% of individuals undergo genetic testing. Furthermore, racial, ethnic, and linguistic minorities experience even greater under-recognition of familial cancer syndromes.This results in a critical missed opportunity for preventing cancer-associated morbidity and mortality. Obstetric care is a potential window of opportunity for addressing this issue, as pregnancy offers a unique opportunity for individuals to interact with the healthcare system. Importantly, patients are already being introduced to the topics of genetic testing and counseling, as the American College of Obstetricians and Gynecologists (ACOG) recommends that all pregnant women receive information regarding carrier screening. The uptake of OCS to evaluate hundreds of disorders is increasing rapidly, with a recent meta-analysis finding that 39% of patients undergo such testing. Currently, however, most cancer-associated mutations are not included in OCS assays. Screening reproductive-age women presents a unique opportunity to perform testing at a time when precancer screening, chemoprevention, and/or risk-reducing surgery is most beneficial.

Limited prior literature suggests that 50-75% of patients would accept combined HCS/OCS if offered. The investigators offered hereditary cancer risk assessment to 100 obstetrical patients in a diverse, Medicaid-predominant Weill Cornell Medicine clinic and found that 66% of patients were interested in cancer risk assessment during pregnancy. Furthermore, the investigators recently published a cost-effectiveness analysis suggesting that incorporation of BRCA1 genetic testing to all patients, regardless of family history at the time of OCS, is a cost-effective management strategy that can result in the prevention of breast and ovarian cancer cases and cancer deaths. Additionally, patient interviews suggest that more than 50% of patients mistakenly believed their OCS included cancer genes. This misconception poses a significant risk, as these patients assume that they had comprehensive testing and no hereditary cancer risk. Therefore, additional testing was believed to be unnecessary. Finally, prior theoretical patient surveys suggest high levels of interest in this combination testing among ethnically diverse populations. However, there has yet to be a prospective study offering patients the combined HCS/OCS, and all reported interests remain theoretical.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years - 55 years
* Pregnant patients receiving obstetrical-related care or receiving preconception/fertility care at a WCM-affiliated enrollment site.
* Patients who have elected to undergo OCS with the WCM-affiliated obstetrics provider
* Patients with prior OCS but planned to repeat OCS are eligible
* Patients can speak and read in English or Spanish

Exclusion Criteria:

* Patients who have previously completed a multigene hereditary cancer syndrome panel
* Patients who have a hematologic cancer or hematologic pre-cancer
* Patients who have a history of an autologous bone marrow transplant

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 550 (Estimated)
Dates: Start 2025-09-02 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants Who Complete Both HCS and OCS | Approximately within the end of recruitment expected at 2 years
  Percentage of enrolled participants who successfully complete both HCS and OCS during the study period. Completion is defined as having documented results for both screenings

SECONDARY OUTCOMES:
Percentage of Participants Completing Both HCS and OCS, Stratified by Demographic and Clinical Characteristics | Approximately at the end of recruitment, expected at 2 years.
  The percentage of participants who complete both HCS and OCS, stratified by patient race, ethnicity, language, gestational age, insurance provider, personal cancer history, and family cancer history. Completion is defined as having documented results for both screenings.
Percentage of High-Risk Participants Utilizing Guideline-Based Cancer Mitigation Strategies | From completion of screening up to 18 months post-screening
  Among participants who complete both HCS and OCS and are identified as being at elevated cancer risk, this measure captures the percentage who undergo one or more guideline-based cancer mitigation strategies, such as mammogram, breast MRI, or colonoscopy.
Participant Experience with Combined HCS and OCS measured by the NCCN Distress Thermometer | The questionnaire is received right after genetic counseling regarding HCS has been received.
  Participant experience with combined HCS and OCS will be assessed using a National Comprehensive Cancer Network (NCCN) validated scale called the Distress Thermometer. It is a single-item scale ranging from 0 (no distress) to 10 (extreme distress). A lower score indicates less distress, while a higher score signifies greater distress.
Participant Experience with Combined HCS and OCS measured by Satisfaction with Genetic Counseling Scale | The questionnaire is received right after genetic counseling regarding HCS has been received.
  Participant experience with combined HCS and OCS will be assessed using a validated Satisfaction with Genetic Counseling Scale. It is a 10-item Likert scale (1-5) assessing satisfaction with counseling, including both positively and negatively worded items (reverse-scored). Total scores range from 10 to 50, with higher scores indicating greater satisfaction.
Participant Experience with Combined HCS and OCS measured by Satisfaction with Decision Scale | The questionnaire is received right after genetic counseling regarding HCS has been received.
  Participant experience with combined HCS and OCS will be assessed using a validated Satisfaction with Decision Scale. It is a 6-item Likert scale (1-5) measuring satisfaction with the decision to undergo genetic testing. Scores range from 6 to 30; higher scores indicate greater satisfaction.
Participant Experience with Combined HCS and OCS - Qualitative Interview | From completion of screening up to 18 months post-screening
  A subset of participants will complete a semi-structured interview to explore their experiences with being offered hereditary cancer screening alongside obstetrical carrier screening. Interview topics include perceptions of how screening information was presented, reasons for accepting or declining genetic testing, challenges faced in the decision-making and testing process, and suggestions for improving the patient experience. Interviews will be audio-recorded with consent, transcribed, and analyzed using thematic analysis.
Provider Experience with Combined HCS and OCS - Qualitative Interview | From completion of screening up to 18 months post-screening
  This qualitative outcome measure assesses providers' experiences with the implementation and delivery of combined HCS and OCS through a semi-structured interview. Themes explored include prior experiences discussing genetic testing during obstetrical visits, perceptions of screening timing and appropriateness during pregnancy, challenges encountered, and suggestions for improving the screening process. Interviews will be audio-recorded, transcribed, and thematically analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Frey, MD, MS, Principal Investigator — Weill Medical College of Cornell University
Locations (5):
- United States (5):
  - Reproductive Medicine, Brooklyn, New York
  - NewYork-Presbyterian Weill Cornell Medicine, Brooklyn, New York
  - Reproductive Medicine, New York, New York
  - Weill Cornell Medicine, New York, New York
  - NewYork-Presbyterian Weill Cornell Medicine Queens, Queens, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Palinkas LA, Horwitz SM, Green CA, Wisdom JP, Duan N, Hoagwood K. Purposeful Sampling for Qualitative Data Collection and Analysis in Mixed Method Implementation Research. Adm Policy Ment Health. 2015 Sep;42(5):533-44. doi: 10.1007/s10488-013-0528-y. PMID 24193818
- [Background] Kaphingst KA, Bather JR, Daly BM, Chavez-Yenter D, Vega A, Kohlmann WK. Interest in Cancer Predisposition Testing and Carrier Screening Offered as Part of Routine Healthcare Among an Ethnically Diverse Sample of Young Women. Front Genet. 2022 Apr 14;13:866062. doi: 10.3389/fgene.2022.866062. eCollection 2022. PMID 35495140
- [Background] Dioun SM, Perez LR, Prabhu M, Brewer JT, Ahsan MD, Hou JY, Sharaf RN, Wright JD, Frey MK. Cost-effectiveness of BRCA1 testing at time of obstetrical prenatal carrier screening for cancer prevention. Am J Obstet Gynecol. 2024 Sep;231(3):330.e1-330.e14. doi: 10.1016/j.ajog.2024.04.014. Epub 2024 Apr 14. PMID 38621481
- [Background] Grant BJ, Chandler I, Son M, Dioun S, Mcdougale A, Sharaf RN, Frey MK. Pregnancy: an underutilized window of opportunity for genetic cancer risk assessment. Am J Obstet Gynecol. 2025 Jan;232(1):e11-e13. doi: 10.1016/j.ajog.2024.09.100. Epub 2024 Sep 19. No abstract available. PMID 39306315
- [Background] Zhong L, Bather JR, Daly BM, Kohlmann WK, Goodman MS, Rothwell E, Kaphingst KA. Investigation of interest in and timing preference for cancer predisposition testing and expanded carrier screening among women of reproductive age. PEC Innov. 2023 Jan 24;2:100128. doi: 10.1016/j.pecinn.2023.100128. eCollection 2023 Dec. PMID 37214524
- [Background] Edwards JG, Feldman G, Goldberg J, Gregg AR, Norton ME, Rose NC, Schneider A, Stoll K, Wapner R, Watson MS. Expanded carrier screening in reproductive medicine-points to consider: a joint statement of the American College of Medical Genetics and Genomics, American College of Obstetricians and Gynecologists, National Society of Genetic Counselors, Perinatal Quality Foundation, and Society for Maternal-Fetal Medicine. Obstet Gynecol. 2015 Mar;125(3):653-662. doi: 10.1097/AOG.0000000000000666. PMID 25730230
- [Background] Goldberg JD, Pierson S, Johansen Taber K. Expanded carrier screening: What conditions should we screen for? Prenat Diagn. 2023 Apr;43(4):496-505. doi: 10.1002/pd.6306. Epub 2023 Jan 18. PMID 36624552
- [Background] Committee Opinion No. 691: Carrier Screening for Genetic Conditions. Obstet Gynecol. 2017 Mar;129(3):e41-e55. doi: 10.1097/AOG.0000000000001952. PMID 28225426
- [Background] ACOG Committee Opinion No. 752: Prenatal and Perinatal Human Immunodeficiency Virus Testing. Obstet Gynecol. 2018 Sep;132(3):e138-e142. doi: 10.1097/AOG.0000000000002825. PMID 30134428
- [Background] Pazol K, Robbins CL, Black LI, Ahrens KA, Daniels K, Chandra A, Vahratian A, Gavin LE. Receipt of Selected Preventive Health Services for Women and Men of Reproductive Age - United States, 2011-2013. MMWR Surveill Summ. 2017 Oct 27;66(20):1-31. doi: 10.15585/mmwr.ss6620a1. PMID 29073129
- [Background] Lin J, Sharaf RN, Saganty R, Ahsan D, Feit J, Khoury A, Bergeron H, Chapman-Davis E, Cantillo E, Holcomb K, Blank SV, Liu Y, Thomas C, Christos PJ, Wright DN, Lipkin S, Offit K, Frey MK. Achieving universal genetic assessment for women with ovarian cancer: Are we there yet? A systematic review and meta-analysis. Gynecol Oncol. 2021 Aug;162(2):506-516. doi: 10.1016/j.ygyno.2021.05.011. Epub 2021 May 19. PMID 34023131
- [Background] Guzauskas GF, Garbett S, Zhou Z, Schildcrout JS, Graves JA, Williams MS, Hao J, Jones LK, Spencer SJ, Jiang S, Veenstra DL, Peterson JF. Population Genomic Screening for Three Common Hereditary Conditions : A Cost-Effectiveness Analysis. Ann Intern Med. 2023 May;176(5):585-595. doi: 10.7326/M22-0846. Epub 2023 May 9. PMID 37155986
- [Background] Offit K. The future of clinical cancer genomics. Semin Oncol. 2016 Oct;43(5):615-622. doi: 10.1053/j.seminoncol.2016.10.002. Epub 2016 Oct 18. PMID 27899195
- [Background] Gabai-Kapara E, Lahad A, Kaufman B, Friedman E, Segev S, Renbaum P, Beeri R, Gal M, Grinshpun-Cohen J, Djemal K, Mandell JB, Lee MK, Beller U, Catane R, King MC, Levy-Lahad E. Population-based screening for breast and ovarian cancer risk due to BRCA1 and BRCA2. Proc Natl Acad Sci U S A. 2014 Sep 30;111(39):14205-10. doi: 10.1073/pnas.1415979111. Epub 2014 Sep 5. PMID 25192939
- [Background] Mandelker D, Zhang L, Kemel Y, Stadler ZK, Joseph V, Zehir A, Pradhan N, Arnold A, Walsh MF, Li Y, Balakrishnan AR, Syed A, Prasad M, Nafa K, Carlo MI, Cadoo KA, Sheehan M, Fleischut MH, Salo-Mullen E, Trottier M, Lipkin SM, Lincoln A, Mukherjee S, Ravichandran V, Cambria R, Galle J, Abida W, Arcila ME, Benayed R, Shah R, Yu K, Bajorin DF, Coleman JA, Leach SD, Lowery MA, Garcia-Aguilar J, Kantoff PW, Sawyers CL, Dickler MN, Saltz L, Motzer RJ, O'Reilly EM, Scher HI, Baselga J, Klimstra DS, Solit DB, Hyman DM, Berger MF, Ladanyi M, Robson ME, Offit K. Mutation Detection in Patients With Advanced Cancer by Universal Sequencing of Cancer-Related Genes in Tumor and Normal DNA vs Guideline-Based Germline Testing. JAMA. 2017 Sep 5;318(9):825-835. doi: 10.1001/jama.2017.11137. PMID 28873162
- [Background] Childers CP, Childers KK, Maggard-Gibbons M, Macinko J. National Estimates of Genetic Testing in Women With a History of Breast or Ovarian Cancer. J Clin Oncol. 2017 Dec 1;35(34):3800-3806. doi: 10.1200/JCO.2017.73.6314. Epub 2017 Aug 18. PMID 28820644
- [Background] US Preventive Services Task Force; Owens DK, Davidson KW, Krist AH, Barry MJ, Cabana M, Caughey AB, Doubeni CA, Epling JW Jr, Kubik M, Landefeld CS, Mangione CM, Pbert L, Silverstein M, Simon MA, Tseng CW, Wong JB. Risk Assessment, Genetic Counseling, and Genetic Testing for BRCA-Related Cancer: US Preventive Services Task Force Recommendation Statement. JAMA. 2019 Aug 20;322(7):652-665. doi: 10.1001/jama.2019.10987. PMID 31429903
- [Background] de Jong AE, Hendriks YM, Kleibeuker JH, de Boer SY, Cats A, Griffioen G, Nagengast FM, Nelis FG, Rookus MA, Vasen HF. Decrease in mortality in Lynch syndrome families because of surveillance. Gastroenterology. 2006 Mar;130(3):665-71. doi: 10.1053/j.gastro.2005.11.032. PMID 16530507
- [Background] Domchek SM, Friebel TM, Singer CF, Evans DG, Lynch HT, Isaacs C, Garber JE, Neuhausen SL, Matloff E, Eeles R, Pichert G, Van t'veer L, Tung N, Weitzel JN, Couch FJ, Rubinstein WS, Ganz PA, Daly MB, Olopade OI, Tomlinson G, Schildkraut J, Blum JL, Rebbeck TR. Association of risk-reducing surgery in BRCA1 or BRCA2 mutation carriers with cancer risk and mortality. JAMA. 2010 Sep 1;304(9):967-75. doi: 10.1001/jama.2010.1237. PMID 20810374
- [Background] Offit K, Tkachuk KA, Stadler ZK, Walsh MF, Diaz-Zabala H, Levin JD, Steinsnyder Z, Ravichandran V, Sharaf RN, Frey MK, Lipkin SM, Robson ME, Hamilton JG, Vijai J, Mukherjee S. Cascading After Peridiagnostic Cancer Genetic Testing: An Alternative to Population-Based Screening. J Clin Oncol. 2020 May 1;38(13):1398-1408. doi: 10.1200/JCO.19.02010. Epub 2020 Jan 10. PMID 31922925